CLINICAL TRIAL: NCT05141097
Title: Quality of Life for Patients Who Are Treated Using Integrative Medicine
Brief Title: Integrative Medicine Quality of Life Study
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ambereen Ahmed, Integrative Medicine Fellow and Junior Faculty, University of Arizona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aahmed2
Record Dates: First submitted 2021-11-06; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Integrative Medicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Being cared for by an Integrative Medicine provider
  Interventions: Other: Integrative medicine approach
- Control (No Intervention): Being cared for by conventional medicine provider

INTERVENTIONS:
Other: Integrative medicine approach — By treated by integrative medicine approaches instead of conventional medicine
  Arms: Treatment

SUMMARY:
Integrative Medicine is an approach to health that addresses a person's mental, physical, social, spiritual, and environmental factors. Chronic diseases are best treated if the root cause is addressed, improving one's overall health. Health is defined by the WHO as "a state of complete physical, mental and social wellbeing, and not merely the absence of disease or infirmity." Many national institutions, such as the American Heart Association, American College of Cardiology, American Diabetes Association, and more, all affirm that lifestyle modifications are the number one treatment and prevention for the most common disorders: high blood pressure, obesity, diabetes, high cholesterol, etc. The generic term "lifestyle modifications" encompasses many aspects that can be impacted by Integrative Medicine.

Patients present to be treated by Integrative Medicine practitioners frequently, and we would like to see how their quality of life is improving by being treated by this practice approach.

DETAILED DESCRIPTION:
At the turn of the 19th century, medicine made great strides in the field of bacteriology. Development of antibiotics, pasteurization, sterilization and antiseptic techniques led to tremendous advances in the understanding of disease pathophysiology.

Unfortunately, with increased longevity came increased rates of chronic diseases, a shift referred to as the "epidemiological transition." Lifestyle risk factors have been directly linked to the increase in diseases, such as heart disease, cancer, and stroke - with these conditions overtaking infectious diseases such as TB, influenza, cholera, and pneumonia as the major sources of mortality in the developed countries.

These major external or modifiable factors contributing to US mortality were subsequently labeled the "actual causes of death" and included tobacco usage, physical inactivity, diet, alcohol, sexual behaviors, and others (McGinnis, 1993). This same analysis has persisted into the 21st century. An analysis by Mokdad published in JAMA, 2004 found that tobacco, poor diet, physical inactivity and alcohol use were the leading causes of death, collectively accounting for 36.8% of all deaths in 2000. In 2014, chronic diseases remain the leading cause of mortality and morbidity in the US and the main contributors to these diseases are tobacco use, poor diet, physical inactivity, alcohol use, hypertension and hyperlipidemia - all modifiable risk factors. As medical research shifted toward addressing these chronic health conditions linked to lifestyle risk factors, the clinical practice of medicine shifted to a disease-oriented model.

At the core of Integrative Medicine, physicia strive to delineate factors that have caused a person to be who they are at this current stage, all the way from when they were in utero until now.

Integrative Medicine is a practice approach to medicine that strives to achieve health, the definition of health being a state of complete physical, mental and social wellbeing, and not merely the absence of disease or infirmity, as defined by the WHO.

The Andrew Weil Center of Integrative Medicine has the following principals at the core of its practice: the patient and practitioner are partners in the healing process; all factors that influence health, wellness and disease are taken into consideration, including mind, spirit and community, as well as the body. Appropriate use of both conventional and alternative methods facilitates the body's innate healing response. Effective interventions that are natural and less invasive should be used whenever possible; the broader concepts of health promotion and prevention of illness are paramount.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are any healthy or non-healthy adult or child
* English-speaking
* Any ethnic background
* Any socioeconomic status

Exclusion Criteria:

* Pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Medical Symptoms Questionnaire | through study completion, anticipated 6 months
  Quantitative review of systems survey, with a maximum score of 280 indicating severe toxicity, and a minimum score of 0 indicating no toxicity. The score breakdown is as following: <10 optimal health, 10-50 mild toxicity, 50-100 moderate toxicity, >100 severe toxicity.
PROMIS Global Health Scale | through study completion, anticipated 6 months
  Qualitative quality of life survey, with a maximum score of 45 indicating great subjective quality of life, and minimum score of 0 indicating very poor subjective quality of life.

IPD SHARING:
Plan to Share IPD: No